CLINICAL TRIAL: NCT02761421
Title: Effect of Motor Development, Motor Function and Electrodiagnostic Characteristic of IOPD Under ERT
Brief Title: Effect of Motor Development, Motor Function and Electrophysiologic Findings of IOPD Under ERT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015-12-014C
Record Dates: First submitted 2016-04-26; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2015-12

CONDITIONS: Glycogen Storage Disease Type II
Keywords: IOPD
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Observational Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with IOPD: observation all patients with IOPD
  Interventions: Other: observation study

INTERVENTIONS:
Other: observation study — observation study

SUMMARY:
To investigate the motor development, motor function and electrodiagnostics presentation in IOPD under ERT.

DETAILED DESCRIPTION:
Background

Pompe disease is an autosomal recessive disease, enzyme replacement therapy (ERT) and new born screen (NBS) had been initiated in Taiwan since 2008. However, residual muscle weakness were noted. Decrease in amplitude of nerve compound muscle action potential (CMAP) and increase spontaneous activity were reported before the imitation of ERT. However, the motor development, motor function and electrodiagnostic presentation which were important in further direction of treatment and rehabilitation program arrangement in infantile Pompe disease (IOPD) under ERT is lacking.

Aim

To investigate the motor development, motor function and electrodiagnostic presentation in IOPD under ERT.

Method

This is an observational, prospective, longitudinal, follow-up study. Motor development was assessed by Alberta Infant Motor Scale (AIMS) and Peabody Developmental Motor Scales, Second Edition (PDMS II); motor function was assessed by Pediatric Evaluation of Disability Inventory (PEDI) and Gross Motor Function Measure (GMFM). Electrodiagnosis studies include nerve conduction study (NCS) and electromyography (EMG).

Expect Effects

Obtain the characteristics of motor development, motor function and electrodiagnosis presentation of IOPD under ERT, and the relation between motor development, motor function and electrodiagnosis presentation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with infantile onset Pompe disease (IOPD) who were diagnosed and follow-up at Taipei Veteran General Hospital (TVGH).

Exclusion Criteria:

* Patients whose guardian did not provide the inform consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators included all patients with infantile onset Pompe disease (IOPD) who were diagnosed and follow-up at Taipei Veteran General Hospital (TVGH) and excluded patients whose guardian did not provide the inform consent.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Raw Score of Alberta Infant Motor Scale Development quotient of Peabody Developmental Motor Scales, Second Edition | 1 year
Development Quotient of PDMS-II | 1 year

SECONDARY OUTCOMES:
Raw Score of Pediatric Evaluation of Disability Inventory Total score of GMFM | 1 year
Total Score of GMFM | 1 year

OTHER OUTCOMES:
Percentile of active denervation in electrodiagnostic study | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veteran General Hospital : Taipei City, Taiwan 11217, R.O.C., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
publication in journal